CLINICAL TRIAL: NCT06667414
Title: Frequency of Selected Single Nucleotide Polymorphisms in Phase With the Mutant and Wild-Type HTT Alleles in Huntington Disease Gene Expansion Carriers
Brief Title: Frequency of Selected Single Nucleotide Polymorphisms in Huntington Disease Gene Expansion Carriers
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: WE45491
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Who Are Huntington Disease Gene Expansion Carriers

SUMMARY:
For participation in this epidemiological study, a single-day visit at the study site is required. Participants will be recruited from Huntington Disease clinics, and they will be asked to answer questions regarding their demographics, including sex, age, race and ethnicity, and their medical and medication history. At the end of the visit, a blood sample will be drawn to allow testing with a sequencing assay that is specifically designed for phasing single nucleotide polymorphisms (SNPs) on the wild-type Huntington (wtHTT) and mutant Huntington (mHTT) alleles.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the Informed Consent Form (ICF)
* Aged 25 to 60 years, inclusive, at the time of signing the ICF
* Confirmation of Huntington Disease (HD) gene expansion mutation carrier status
* Confirmation of Total Functional Capacity (TFC) ≥9 and Total Motor Score (TMS) >6 within 12 months prior to signing the ICF
* Ability to tolerate blood draws

Exclusion Criteria:

* None

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This epidemiological study will be conducted in ambulatory men and women aged 25 to 60 years old (inclusive) who carry the Huntington Disease (HD) gene expansion and meet the Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score (TMS) and Total Functional Capacity (TFC) criteria for HD Integrated Staging System (HD-ISS) Stages 2-3.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2028-09-24 (Estimated); Study Completion 2028-09-24 (Estimated)

PRIMARY OUTCOMES:
Frequencies of Selected Single Nucleotide Polymorphism (SNP) Alleles in Phase With the mHTT and wtHTT Alleles | Day 1

SECONDARY OUTCOMES:
Number of Participants With Selected SNPs According to Their Medical History | Day 1
Number of Participants With Selected SNPs According to Their Medication History | Day 1
Number of Participants With Selected SNPs According to Their Demographic Characteristics (Age, Sex, Ethnicity, and Race) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (13):
  - Uab Medicine, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - University of California Davis Medical System, Sacramento, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - EvergreenHealth Investigational Drug Services, Kirkland, Washington
- Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires, Argentina
- Australia (4):
  - Calvary Health Care Bethlehem, Caulfield South, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Melbourne Hospital, Parkville, Victoria
  - Graylands Hospital, Mount Claremont, Western Australia
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Centricity Research, Halifax, Nova Scotia
  - North York General Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- Rigshospitalet, Hukommelsesklinikken, København Ø, Denmark
- Germany (4):
  - Charité - Universitätsmed. Berlin, Klinik für Psychiatrie und Psychotherapie, Berlin
  - St. Josef-Hospital, Neurologische Klinik der Ruhr-Uni, Bochum
  - Universitätsklinikum Erlangen, Abteilung Molekulare Neurologie, Erlangen
  - Universitätsklinikum Ulm, Ulm
- Italy (2):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Universita Degli Studi Di Firenze, Florence, Tuscany
- New Zealand (3):
  - Auckland DHB - Neurlogy Department, Auckland
  - New Zealand Brain Research Institute, Christchurch
  - Wellington Hospital, Wellington
- Poland (2):
  - Szpital Sw. Wojciecha, Gda?sk
  - Wojskowy Instytut Medycyny Lotniczej, Warsaw
- Portugal (2):
  - Unidade Local de Saude de Santa Maria, E.P.E. - Hospital de Santa Maria, Lisbon
  - CNS - Campus Neurológico, Torres Vedras
- Spain (4):
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos. Servicio de Neurología, Burgos
  - Hospital Ramon y Cajal, Madrid
- United Kingdom (4):
  - Birmingham and Solihull Mental Health Foundation NHS Trust, Birmingham
  - Addenbrookes Hospital, Cambridge
  - National Hospital For Neurology and Neurosurgery, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No